CLINICAL TRIAL: NCT05958732
Title: Effect of Body Awarness Therapy on Balance and Coordination in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 0352-22
Record Dates: First submitted 2023-05-09; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: Stroke; Balance,; Coordination; mini-mental scale; BBS; Cognition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Experimental group will be receiving conventional therapy and body awareness therapy for 30 minutes, 5 days a week for two weeks. Balance and coordination is measured before the treatment and after two weeks of treatment session it is again measured.
  control group will receive conventional physical therapy treatment for 30 minutes, 5 days a week for two weeks. Balance and coordination is measured before the treatment and after two weeks of treatment session it is again measured.
Who Masked: Participant
Masking Description: The participants will be masked for the treatment groups. Non of the participants know to which treatment group they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive body awareness therapy for 20 minutes.The following steps will be conducted, (1) Put your left hand on your right toe. (2) Put your right hand on your left toe. (3) Touch your heels. (4) Put your feet together. (5) Put your knees together. (6) Touch your right knee with your left hand. (7) Touch your left knee with your right hand. (8) Touch one knee and one foot. (9) Put your right hand on your left knee. (10) Put your left hand on your right knee. (11) Put your feet apart. (12) Touch your toes with your arms crossed. (13) Touch your thumbs to your toes. (14) Bend your knees. (15) Stamp your feet. Duration is 5 days a week for two weeks. Along with conventional therapy.
  Interventions: Other: Somato-sensorial exercises therapy; Other: Conventional Therapy
- Control group (Other): conventional training plan: (1) 5 minute warm up then, (2) static balance exercises, such as, Two leg stance, One Leg stance, and (3) dynamic balance exercises such as, sideway walking with crossover, Forward walking or running in a zigzag line, Backward walking or running in a zigzag line, Jogging end to end, (4) Coordination exercises such as, Tandem stepping, Finger to nose, Finger to finger, Sitting with Shifting weight in all directions, Rebound Phenomenon and cool down for 5 minutes.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Somato-sensorial exercises therapy — It includes exercises, which is already mentioned in the arm description.
  Arms: Experimental Group
Other: Conventional Therapy — It Includes routine exercises for the stroke patient the detail is already given in the arm description.

SUMMARY:
Stroke is sudden disruption in central nervous system function due to disturbance of the blood flow circulation in the brain. Cerebrovascular accident (CVA), is the second most leading cause of mortality (5.5 million cases yearly). Its occurrence remains high, with 13.7 million annual incident cases globally. Ischemic strokes are more common with a prevalence ratio of 76-119 per 100,000 per year worldwide ). Stroke is a neurological disease that decrease sensorimotor functions by causing irreversible impairments to the nervous system due to cerebral vascular problems . Patients with balance and activity disturbance are indicated by reduce in body functions. It is very essential for CVA patients to improve balance stability and muscle power for recovery and for normal activities ). Balance is an essential factor for independent living. It is maintained by adjusting COG (Center of Gravity) over the BOS (Base of Support). These adjustments are done through sensational inputs from the vestibular, visual and somatosensory system and are maintained by brain.

DETAILED DESCRIPTION:
Impairment of balance stability is common in stroke patients. Patients with cerebrovascular accident (CVA) present mainly with asymmetric standing balance that affects their stability limits, and leads to major difficulty in functional independence. A reduction in maintaining balance is one of the major element that adversely affect after stroke. Coordination is another important factor, which allows a person to perform purposeful movement. After cerebrovascular accidents mainly impairment in coordination may be an element in mobility and movement limitations. Restoring the coordinated movement after cerebrovascular accident in important in regaining normal living activities. Those patients who survive from stroke may experience instant changes in thinking, language, balance, coordination, proprioception, body functions and quality of life. Stroke rehabilitation is the restoring functions of the impaired body regions and it is a long and time taking process, both for patients and for rehabilitation teams. Body awareness therapy (BAT) is a physiotherapeutic restorative approach that examine the patient's condition and focus towards relearning self-awareness movements. Body awareness therapy helps in strengthening the patient and also performing in activities of daily living (ADLs). A basic movement is stimulation of center line by weight shifting from right towards left and rotatory movements around the center of body and vice versa. Movements can be achieved in supine, sitting and standing position. Unfortunately, no randomized controlled trial (RCT) study has so far evaluated the effect of body awareness therapy (BAT) on balance and coordination in stroke survivals. Therefore, the purpose of this study is to assess BAT on balance and coordination in patients with cerebrovascular accident (CVA).

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female gender.
2. Sub-acute hemiplegic stroke patients.
3. Age 30 or older.

Exclusion Criteria:

1. Other comorbid conditions.
2. Neurological diseases other than stroke are excluded
3. Severe cognitive impairment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-07-25 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Balance | 2 weeks
  The assessment tests need individual corporation and the assessment is about 15 to 20 minutes. Berg Balance Scale involves 14 different tasks that can be categorized into different domains. Each task is divided into five grades for assessing the level of stability and un-stability and grades are from zero to four. Zero is graded when the person is unable and not performing the task fully and four is given when the person is fully able and able to perform the task independently. However, the score of the Berg balance scale ranges from 0 to 56. The score can be calculated or measured after assessment. From zero to twenty (0-20) severe impairment. From score Twenty-one to forty (21-40) moderate impairment. From score forty-one to fifty-six (41-56) minimal impairment.
Co-ordination | 2 weeks
  The tests that can be performed to measure the coordination of the upper region and the lower region can be equilibrium and non-equilibrium tests.
  The non-Equilibrium test is a simple and very effective clinical assessment screening test and would be assessed as the Finger nose test, Finger Finger Test, and Rebound Phenomena. For the lower limb heel-to-shin test, draw a circle test.
  Equilibrium tests can be performed in a sitting position, in a standing position, and in a walking position. Coordination tests whether equilibrium or non-equilibrium can be assessed into five grades from 0 grade to 4 grade. Grade 0 (Activity Impossible) Grade 1 (severe Impairment) Grade 2 (moderate Impairment) Grade 3 (Minimal Impairment) Grade 4 ( normal Performance).
Cognition | 2 weeks.
  The Mini-Mental State examination is used to check cognition, and orientation, registration, attention and calculation, and memory recall of the objects. The score of the mini-mental state examination ranges between 0 to 30. If the score ranges between thirty to twenty-four (30 to 24) then there is no cognitive impairment. If the score ranges between twenty-three to eighteen (23 to 18) then there is mild cognitive impairment. If the score ranges between seventeen to zero (17-0) then an individual is suffering from severe cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Roshneck Haneed, MS-PT*, Principal Investigator — Shifa Tameer-e-Millat University
Locations (1):
- Shifa Tameer-e-Millat University Islamabad, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang DH, Cho HS. Effect of body awareness training on balance and walking ability in chronic stroke patients: a randomized controlled trial. J Phys Ther Sci. 2016 Jan;28(1):198-201. doi: 10.1589/jpts.2016.198. Epub 2016 Jan 30. PMID 26957757
- [Background] Barclay RE, Stevenson TJ, Poluha W, Semenko B, Schubert J. Mental practice for treating upper extremity deficits in individuals with hemiparesis after stroke. Cochrane Database Syst Rev. 2020 May 25;5(5):CD005950. doi: 10.1002/14651858.CD005950.pub5. PMID 32449959
- [Background] Choi JU, Kang SH. The effects of patient-centered task-oriented training on balance activities of daily living and self-efficacy following stroke. J Phys Ther Sci. 2015 Sep;27(9):2985-8. doi: 10.1589/jpts.27.2985. Epub 2015 Sep 30. PMID 26504340
- [Background] Doost MY, Orban de Xivry JJ, Herman B, Vanthournhout L, Riga A, Bihin B, Jamart J, Laloux P, Raymackers JM, Vandermeeren Y. Learning a Bimanual Cooperative Skill in Chronic Stroke Under Noninvasive Brain Stimulation: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2019 Jun;33(6):486-498. doi: 10.1177/1545968319847963. Epub 2019 May 15. PMID 31088342
- [Background] Kass B, Dornquast C, Meisel A, Holmberg C, Rieckmann N, Reinhold T. Cost-effectiveness of patient navigation programs for stroke patients-A systematic review. PLoS One. 2021 Oct 15;16(10):e0258582. doi: 10.1371/journal.pone.0258582. eCollection 2021. PMID 34653188
- [Background] Kim JC, Lim JH. The effects of coordinative locomotor training on coordination and gait in chronic stroke patients: a randomized controlled pilot trial. J Exerc Rehabil. 2018 Dec 27;14(6):1010-1016. doi: 10.12965/jer.1836386.193. eCollection 2018 Dec. PMID 30656163
- [Background] Kutlay S, Genc A, Gok H, Oztuna D, Kucukdeveci AA. Kinaesthetic ability training improves unilateral neglect and functional outcome in patients with stroke: A randomized control trial. J Rehabil Med. 2018 Feb 13;50(2):159-164. doi: 10.2340/16501977-2301. PMID 29209731
- [Background] Lindvall MA, Anderzen Carlsson A, Forsberg A. Basic Body Awareness Therapy for patients with stroke: Experiences among participating patients and physiotherapists. J Bodyw Mov Ther. 2016 Jan;20(1):83-89. doi: 10.1016/j.jbmt.2015.06.004. Epub 2015 Jun 15. PMID 26891641
- [Background] Yoo J, Jeong J, Lee W. The effect of trunk stabilization exercise using an unstable surface on the abdominal muscle structure and balance of stroke patients. J Phys Ther Sci. 2014 Jun;26(6):857-9. doi: 10.1589/jpts.26.857. Epub 2014 Jun 30. PMID 25013283